CLINICAL TRIAL: NCT03648905
Title: Clinical Laboratory Evaluation of Chronic Autonomic Failure
Status: Active, not recruiting | Type: Observational
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 180140; 18-N-0140
Record Dates: First submitted 2018-08-24; First posted 2018-08-28 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01-20

CONDITIONS: Parkinson's Disease; Multiple System Atrophy; Autonomic Failure
Keywords: Autonomic Failure; Parkinson's Disease; Multiple System Atrophy; Lewy Body; Catecholamines
MeSH Terms: conditions — Parkinson Disease; Multiple System Atrophy; Pure Autonomic Failure | interventions — fluorodopa F 18

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Control patients (iatrogenic CAF): Patients with iatrogenic chronic autonomic failure (CAF) (e.g., status-post cardiac transplantation, pre/post bilateral thoracic sympathectomies)
  Interventions: Drug: 13N-Ammonia; Drug: 18F-DOPA; Drug: 11C-Methylreboxetine (11C-MRB); Drug: 18F-Dopamine
- Control patients (PD No OH): Patients with Parkinson's disease (PD) without orthostatic hypotension (PD no OH)
  Interventions: Drug: 13N-Ammonia; Drug: 18F-DOPA; Drug: 11C-Methylreboxetine (11C-MRB); Drug: 18F-Dopamine
- Healthy Volunteers: Healthy Volunteers, includes people with genetic risk of PD or studied as concurrent controls
  Interventions: Drug: 13N-Ammonia; Drug: 18F-DOPA; Drug: 11C-Methylreboxetine (11C-MRB); Drug: 18F-Dopamine
- Patients with neurodegenerative chronic autonomic failure (CAF): Includes patients with orthostatic hypotension (OH) due to sympathetic neurocirculatory failure (nOH), and people with multiple system atrophy (MSA).
  Interventions: Drug: 13N-Ammonia; Drug: 18F-DOPA; Drug: 11C-Methylreboxetine (11C-MRB); Drug: 18F-Dopamine

INTERVENTIONS:
Drug: 13N-Ammonia — a perfusion imaging agent
Drug: 18F-DOPA — is a positron-emitting analog of the catechol amino acid, levodopa
Drug: 11C-Methylreboxetine (11C-MRB) — 11C-MRB may be injected IV for visualizingsites of neuronal uptake of norepinephrine in the brain or periphery by PET scanning. Setup includes placement of an arm IV catheter. 11C-MRB is a Radioactive Research Drug.
Drug: 18F-Dopamine — is a positron-emitting analog of the catecholamine, dopamine

SUMMARY:
Background:

The autonomic nervous system controls automatic body functions. Researchers want to improve the tests used to diagnose autonomic failure. Orthostatic hypertension is a drop in blood pressure when a person stands up. Researchers want to focus on this sign of autonomic failure.

Objective:

To improve testing for conditions that cause autonomic nervous system failure.

Eligibility:

People ages 18 and older in one of these categories:

* Their blood pressure drops when they get up.
* They have had a heart transplant or bilateral endoscopic thoracic sympathectomies or have had or will have renal sympathetic ablation

Design:

All participants will be screened with:

* Medical history
* Physical exam
* Blood and urine tests

Some participants will be screened with:

* Heart and breathing tests
* IV placement into an arm vein
* Tilt table testing: Participants lie on a table that tilts while an IV is used to draw their blood.

Participants may stay in the hospital for up to 1 week depending on their tests. Tests may include repeats of screening tests and:

* Sweat testing: A drug is placed on the skin to cause sweating. Sensors on the skin measure moisture.
* Lumbar puncture: A needle is inserted between the bones in the back to collect fluid.
* MRI and PET/CT scan: Participants lie on a table that slides into a scanner. For the PET/CT, a small amount of a radioactive chemical will be injected with a small amount of a radioactive chemical.
* Bladder catheter placement to collect urine
* Skin biopsies: A punch tool removes a small skin sample.
* Tests to see how the pupils react to light
* Smelling tests
* Thinking and memory tests
* Questionnaires

Participants may have a visit about 2 years later to repeat tests.

DETAILED DESCRIPTION:
Objective: In dysautonomias, altered function of one or more components of the autonomic nervous system adversely affect health. A subset of dysautonomias consists of chronic autonomic failure (CAF) syndromes. A key sign of CAF is orthostatic hypotension (OH) due to sympathetic neurocirculatory failure (neurognic OH, or nOH). Primary CAF has been classified based on clinical manifestations into three forms - pure autonomic failure (PAF), multiple system atrophy (MSA), and Parkinson's disease with OH (PD+OH). All three forms involve deposition of the protein alpha-synuclein (AS) in neurons (PD, PAF) or glial cells (MSA), and therefore are called autonomic synucleinopathies. Clinical assessment alone often is inadequate for distinguishing among these conditions in individual patients. This observational study continues and expands on Protocol 03-N-0004, "Clinical Laboratory Evaluation of Primary Chronic Autonomic Failure." The overall objective is to refine and conduct multi-modality testing of catecholaminergic and autonomic systems in patients with CAF. The goals are to: (a) improve the differential diagnosis of CAF via laboratory biomarkers; (b) track the natural history of CAF by follow-up testing; (c) apply clinical laboratory biomarkers to gain insights into underlying pathophysiological mechanisms of CAF; and (d) build up rosters of well characterized patients for future experimental therapeutic trials.

Study Population: The study population consists of patients with neurodegenerative CAF identified by on-site screening at the NIH Clinical Center. Comparison groups include control patients with iatrogenic CAF (e.g., status-post cardiac transplantation, pre/post bilateral thoracic sympathectomies) or PD without OH (PD No OH), and Healthy Volunteers (HVs). MSA patients are included, to build up a subject roster for a planned clinical trial.

Design: This is an observational pathophysiology/natural history study with a planned duration of 5 years. Descriptive statistics will be done in diagnostic groups with neurodegenerative CAF.

Outcome Measures: The study is hypothesis generating/exploratory. The primary outcome measure is results of clinical laboratory research tests. Neurobehavioral rating scales include the University of Pennsylvania Smell Identification Test (UPSIT), Montreal Cognitive Assessment (MoCA), and Uniform Parkinson's Disease Rating Scale (UPDRS). Neurochemical data are from assays of catechols and related compounds in plasma or cerebrospinal fluid. Neuroimaging data are from 18F-DOPA, 18F-dopamine, 13N-ammonia, and 11C-methylreboxetine positron emission tomographic (PET) scanning and MRI. Immunofluorescence microscopy is used to quantify immunoreactive tyrosine hydroxylase and AS in skin biopsy samples. Correlation analyses are done among individual values for outcome measures.

ELIGIBILITY:
* INCLUSION CRITIERIA:

Inclusion Critieria: Patients referred for orthostatic hypotension. This is the main subject cohort.

* Previously studied and diagnosed with one of the forms of nOH or else newly accrued with a referral diagnosis of orthostatic hypotension, and
* 18 years or older, and
* Able to provide own consent to participate or have an existing Legally Authorized Representative (LAR).

If a patient has already been diagnosed as having neurodegenerative CAF under NIH Clinical Protocol 03-N-0004, this satisfies the inclusion criteria for that patient. Previous enrollment in NIH Clinical Protocol 03-N-0004 is not required for enrollment in this study. We do plan to recruit participation into this study from NIH Clinical Protocol 03-N-0004, which has been closed.

If a patient has been referred for OH, then the patient gives consent at the NIH Clinical Center (and therefore is accrued) and then has screening testing at the NIH Clinical Center to confirm that the OH is neurogenic. We anticipate that all patients referred for OH will be shown to have nOH upon screening testing at the NIH Clinical Center. At the time of screening, exclusionary abnormal laboratory test results (e.g., high serum creatinine indicating renal failure) may come to light, in which case they will be withdrawn from the study; however, the patient would have been accrued.

Inclusion criteria: Control patients with iatrogenic CAF

* Patients with heart transplants or pre- or post-bilateral endoscopic thoracic sympathectomies, and
* 18 years or older, and
* Able to provide own consent to participate.

Inclusion criteria: Control patients with PD No OH:

* Patients with PD and no OH who have (a) already been evaluated under other protocols of the AMS and are undergoing follow-up; (b) have already been evaluated under another intramural NINDS protocol; or (c) have cardiac symptoms, signs, or laboratory findings that in the opinion of the PI make it likely there is a cardiac sympathetic lesion, and
* 18 years or older, and
* Able to provide own consent to participate.

Inclusion criteria: Healthy Volunteers:

* Age 18 years or older, and
* Able to provide own consent to participate.

NIH employees may participate. There is no direct solicitation of employees/staff by supervisors. Co-workers will not solicit co-workers. NIH employees are required to abide by NIH Policy Manual 2300-630-3, "Leave Policy for NIH Employees Participating in NIH Medical Research Studies."

EXCLUSION CRITIERIA:

Patient Group Referred for Orthostatic Hypotension

* A medical condition that in the judgment of the Principal Investigator would place the subject at substantially increased acute medical risk, or
* A disqualifying condition such as: hepatic or renal failure, symptomatic congestive heart failure, severe anemia, psychosis, refractory ventricular arrhythmias, currently symptomatic coronary heart disease, cerebrovascular disease with current symptoms (e.g., recent transient ischemic attacks), diabetes, or
* Secondary form of CAF, such as diabetic autonomic neuropathy, or
* Being treated currently (within 2 weeks of anticipated protocol participation) with a medication known to interfere with the cell membrane norepinephrine transporter, which would obviate obtaining scientifically valid results (e.g., tricyclic antidepressant).
* Condition that may cause difficulty or inability to insert a catheter into a vein, or
* Unable to tolerate lying still for up to 1 hour during the procedures, or
* Refusal to undergo certain procedures. These include: (1) IV catheter and blood drawing; (2) DNA extraction, storage, and analysis; (3) PET scanning; or
* Unable to travel safely to the NIH CC, or
* Lacking consent capacity, unless a Durable Power of Attorney (DPA) is in place, or
* Pregnant or breast feeding, or
* Subordinates of study investigators or relatives of the PI or AIs.

Patient Control Group with Iatrogenic CAF or PD No OH

* A medical condition which in the judgment of the Principal Investigator would place the subject at substantially increased acute medical risk, or
* A disqualifying condition such as: hepatic or renal failure, symptomatic congestive heart failure, severe anemia, psychosis, refractory ventricular arrhythmias, currently symptomatic coronary heart disease, cerebrovascular disease with current symptoms (e.g., recent transient ischemic attacks), or diabetes, or
* Being treated currently (within 2 weeks of anticipated protocol participation) with a medication that would obviate obtaining scientifically valid results (e.g., tricyclic antidepressant).
* Condition that may cause difficulty or inability to insert a catheter into a vein, or
* Unable to tolerate lying still for up to 1 hour during the procedures, or
* Refusal to undergo certain procedures. These include: (1) IV catheter and (2) PET scanning, or
* Unable to travel safely to the NIH CC, or
* Lacking consent capacity, or
* Pregnant or breast feeding, or
* Subordinates of study investigators or relatives of the PI or AIs.

Healthy Volunteer Group

* A medical condition which in the judgment of the Principal Investigator would place the subject at substantially increased acute medical risk, or
* A disqualifying condition such as: hepatic or renal failure, symptomatic congestive heart failure, severe anemia, psychosis, refractory ventricular arrhythmias, currently symptomatic coronary heart disease, cerebrovascular disease with current symptoms (e.g., recent transient ischemic attacks), diabetes, or
* Being treated currently (within 2 weeks of anticipated protocol participation) with a medication that would obviate obtaining scientifically valid results (e.g., tricyclic antidepressant).
* Condition that may cause difficulty or inability to insert a catheter into a vein, or
* Unable to tolerate lying still for up to 1 hour during the procedures, or
* Refusal to undergo certain procedures. These include: (1) IV catheter and (2) PET scanning, or
* Unable to travel safely to the NIH CC, or
* Lacking consent capacity, or
* Pregnant or breast feeding, or
* Subordinates of study investigators or relatives of the PI or AIs.

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population consists of patients with neurodegenerative CAF and patients with MSA. Comparison groups include control patients with iatrogenic CAF, patients with PD without OH (PD No OH), and Healthy Volunteers (HVs).
Sampling Method: Non-Probability Sample
Enrollment: 89 (Actual)
Dates: Start 2018-09-06 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Results of clinical laboratory research tests | Initial Visit and on an approximately biennial basis
  Neurobehavioral rating scales include the University of Pennsylvania Smell Identification Test (UPSIT), Montreal Cognitive Assessment (MoCA), and Uniform Parkinson s Disease Rating Scale (UPDRS). Neurochemical data are from assays of catechols and related compounds in plasma or cerebrospinal fluid. Neuroimaging data are from 18F-DOPA, 18Fdopamine, 13Nammonia, and 11Cmethylreboxetine positron emission tomographic (PET) scanning and MRI. Immunofluorescence microscopy is used to quantify immunoreactive tyrosine hydroxylase and AS in skin biopsy samples.

CONTACTS AND LOCATIONS:
Overall Officials: Justin Y Kwan, M.D., Principal Investigator — National Institute of Neurological Disorders and Stroke (NINDS)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2018-N-0140.html